CLINICAL TRIAL: NCT05031858
Title: Effect of Vojta Therapy in Respiratory Disease Caused by SARS-CoV-2. Randomized Controlled Pilot Study
Brief Title: Effect of Vojta Therapy on Covid-19 Respiratory Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NUMEN Foundation (Other)
Collaborators: Hospital de Emergencias Enfermera Isabel Zendal de Madrid (Unknown)
Responsible Party: Principal Investigator, Luis Perales Lopez, Doctor, NUMEN Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Numen3
Record Dates: First submitted 2021-08-28; First posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: COVID-19 Acute Respiratory Distress Syndrome
Keywords: Vojta therapy; Respiratory physiotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vojta Therapy (Experimental): Reflex turn first phase: Patient positioned supine with legs flexed 30º-45º. The pectoral area is stimulated for five minutes on each side x 2 consecutive times. Total 20 minutes per session.
  Interventions: Other: Respiratory physiotherapy
- Control Group (Active Comparator): .Inspiratory techniques, mucociliary clearance techniques (expiratory). Use of inspiratory and expiratory incentives. Employment of mechanical assistants
  Interventions: Other: Respiratory physiotherapy

INTERVENTIONS:
Other: Respiratory physiotherapy — Respiratory physiotherapy

SUMMARY:
Vojta therapy is a physiotherapy intervention with scientific evidence in respiratory pathologies in children and proven in adults. In this pilot study with an RCT design, its effect in adult patients with respiratory pathology caused by the SARS-CoV-2 virus will be studied. The non-invasive and non-painful technique consists of applying tolerable pressure to specific areas of the patient's body. The objective is to activate, in a reflex way, the ventilatory physiology. It is compared with the conventional respiratory physiotherapy approach.

ELIGIBILITY:
Inclusion Criteria:

* respiratory disease by covid-19

Exclusion Criteria:

* patient older than 75 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09-25 (Estimated); Primary Completion 2021-12-20 (Estimated); Study Completion 2022-04-15 (Estimated)

PRIMARY OUTCOMES:
SpO2 | 3 weeks
  Oxygen saturation
Breathing frequency | 3 weeks
  frequency of respiratory cycles per minute
Stay time | 3 weeks
  Days of stay in the intermediate respiratory care unit